CLINICAL TRIAL: NCT00550199
Title: A Phase I Study of LBH589 in Combination With Gemcitabine in the Treatment of Solid Tumors
Brief Title: LBH589 and Gemcitabine in the Treatment of Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to LBH589 toxicity.
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI REFMAL 120; IND 79,355
Record Dates: First submitted 2007-10-26; First posted 2007-10-29 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Solid Tumors
Keywords: Solid Tumors; Phase I; LBH589; Gemcitabine
MeSH Terms: interventions — Panobinostat; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LBH589 and Gemcitabine (Experimental): Phase I dose escalation study
  Interventions: Drug: LBH589, Gemcitabine

INTERVENTIONS:
Drug: LBH589, Gemcitabine — Phase I dose escalation: LBH589 will be administered orally twice weekly. Gemcitabine will be administered intravenously over 30 minutes on days 1, 8, and 15 every 28 days.

SUMMARY:
This will be a single center phase I dose escalation trial. LBH589 will be administered orally twice weekly. Gemcitabine will be administered intravenously over 30 minutes on days 1, 8, and 15 every 28 days. Dose escalation will begin at Dose Level 1. Three patients will be enrolled at each dose level. If 1/3 patients experiences dose-limiting toxicity, the dose level will be expanded to 6 patients. If 2/6 patients experience dose-limiting toxicity at a specific dose level, then the previous dose level will be considered the recommended phase II dose. Dose escalation will continue until the maximum tolerated dose is determined or until all dose levels outlined in the protocol have been completed. A total of 10 patients will be treated at the dose that is recommended for further phase II evaluation to further assess the safety of the combination regimen. Toxicity assessments will be ongoing and disease assessments will be repeated every 2 treatment cycles. Patients will be allowed to continue on study until disease progression unless toxicity warrants drug discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented metastatic or locally advanced, incurable malignancy for which gemcitabine is clinically appropriate (e.g., non-small cell lung cancer, breast, ovarian, bladder cancer and lymphoma).
2. Male or female patients aged ≥ 18 years old.
3. Maximum of 3 prior regimens in a metastatic setting allowed and may include other targeted agents, immunotherapy and chemotherapy.
4. Measurable disease by RECIST criteria.
5. ECOG PS 0 or 1.
6. Laboratory values as follows:

   * ANC > 1500/μL
   * Hgb > 9 g/dL
   * Platelets >100,000/uL
   * Bilirubin < 1.5 mg/dL
   * AST/SGOT and ALT/SGPT < 2.5 x ULN or < 5.0 x ULN in patients with liver metastases
   * Creatinine < 2.0 mg/dL Or 24-hour Creatinine Clearance > 50 ml/min
   * Albumin > 3 g/dL
   * Potassium > lower limit normal (LLN)
   * Phosphorous > LLN
   * Calcium > LLN
   * Magnesium > LLN

8. Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to start of treatment. 9. Life expectancy > 12 weeks. 10. Accessible for treatment and follow-up. 11. All patients must be able to understand the nature of the study and be given written informed consent prior to study entry.

Exclusion Criteria:

1. Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer. Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first LBH589 treatment
2. Impaired cardiac function including any of the following:

   * Screening ECG with a QTc > 450 msec.
   * Congenital long QT syndrome.
   * History of sustained ventricular tachycardia.
   * Any history of ventricular fibrillation or torsades de pointes.
   * Bradycardia defined as heart rate < 50 beats per minutes. Patients wit a pacemaker and heart rate > 50 beats per minute are eligible.
   * Myocardial infarction or unstable angina within 6 months of study entry.
   * Congestive heart failure (NY Heart Association class III or IV.
   * Right bundle branch block and left anterior hemiblock (bifasicular block).
   * Atrial fibrillation or flutter.
3. Uncontrolled hypertension (systolic blood pressure [BP] 180 or diastolic BP >100mm Hg) or uncontrolled cardiac arrhythmias.
4. Active CNS disease, including meningeal metastases.
5. Known diagnosis of human immunodeficiency virus (HIV) infection.
6. Unresolved diarrhea > CTCAE grade 1.
7. Chemotherapy, investigational drug therapy, major surgery < 4 weeks prior to starting study drug or patients that have not recovered from side effects of previous therapy.
8. Patient is < 5 years free of another primary malignancy except if the other primary malignancy is not currently clinically significant or requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
9. Concomitant use of any anti-cancer therapy or radiation therapy other than protocol required gemcitabine.
10. Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not willing to use a double barrier method of contraception during the study and 3 months after the end of treatment. One of these methods of contraception must be a barrier method. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 7 days of the first administration of oral LBH589.
11. Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom.
12. Patients with gastrointestinal (GI) tract disease, causing the inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis).
13. Other concurrent severe, uncontrolled infection or intercurrent illness, including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
14. Patients with uncontrolled coagulopathy.
15. Abnormal thyroid function (TSH or free T4) detected at screening. Patients with known hypothyroidism who are stable on thyroid replacement are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated doses and dose limiting toxicities of LBH589 in combination with gemcitabine when administered to patients with advanced incurable malignant solid tumors. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Howard Burris, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States